CLINICAL TRIAL: NCT05881980
Title: Efficacy and Safety of Terbinafine and Itraconazole Monotherapy in Conventional and Increased Doses and in Combination in Dermatophytosis
Brief Title: Efficacy and Safety of Terbinafine and Itraconazole
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Dr. Afsana Nahid, Assistant professor, Dhaka Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC-DMC/ECC/2023/81
Record Dates: First submitted 2023-05-01; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Tinea Corporis; Tinea Cruris; Tinea Faciei; Dermatophytoses
MeSH Terms: conditions — Tinea; Tinea Cruris | interventions — Terbinafine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group T1 (Experimental): Terbinafine 250 mg/day will be given in this group
  Interventions: Drug: Terbinafine Tablets
- Group I1 (Experimental): Itraconazole 200 mg/day will be given in this group
  Interventions: Drug: Itraconazole
- Group T+I (Experimental): Terbinafine 250 mg + Itraconazole 200 mg/day will be given in this group
  Interventions: Drug: Terbinafine Tablets; Drug: Itraconazole
- Group T2 (Experimental): Terbinafine 500 mg/day in two divided doses will be given in this group
  Interventions: Drug: Terbinafine Tablets
- Group I2 (Experimental): Itraconazole 400 mg/day in two divided doses will be given in this group
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Terbinafine Tablets — Terbinafine 250 mg/day
  Other Names: Terbinafine 250
  Arms: Group T+I; Group T1; Group T2
Drug: Itraconazole — Itraconazole 200 mg/day
  Other Names: Itraconazole 200
  Arms: Group I1; Group I2; Group T+I

SUMMARY:
There is a rise in the prevalence in recent years especially in tropical countries along with an increase in the number of treatment failures with chronic and recurrent dermatophytosis. There is a huge gap between the treatment required in the present scenario and the treatment guidelines given in the standard books. The aim of the study is to determine the effectiveness of terbinafine and itraconazole in different doses and in combination in the treatment of dermatophytosis. The study design will be a randomized parallel-group trial. Patients will be randomly divided into five parallel arms in which two of the standard drugs in recommended doses will be compared with their double doses and with a combination of both drugs. The patients will be reevaluated at 2, 4, 6, and 8 weeks of treatment (the end of therapy), using the physician Global Assessment (PGA) Scale. The cure will be considered a complete clinical resolution of the lesions. The patient's response to the treatment will be recorded. Safety and patient compliance will be recorded at each follow-up visit. Findings of observation will be recorded on a pre-prescribed and pre-tested data collection form. After collection, all data will be checked and compiled. Data will be processed and analyzed using computer software with statistical packages for social science SPSS-26. An analysis plan will be developed keeping in view the objectives of the study. The results of the continuous measurement will be presented on mean ± SD (mean-max) and results on categorical measurements will be presented in numbers (%). A p<0.05 will be considered statistically significant. Results will be disseminated to all Dermatology departments in Bangladesh.

DETAILED DESCRIPTION:
Dermatophyte infections are common fungal infections aggravated by hot and humid climates. Unprecedented changes in the epidemiology, clinical features, and treatment responsiveness of dermatophyte infections have been noted in the recent past in Bangladesh, with many patients presenting with treatment failure and chronic relapsing tinea. Terbinafine and itraconazole are commonly used oral antifungal agents for the same. There is a paucity of original studies especially in Bangladesh depicting dermatophytosis becoming a huge menace both to the patient and to the treating physician. Terbinafine is a fungicidal drug and acts by inhibiting the enzyme squalene epoxidase which converts squalene to lanosterol. Itraconazole is basically a fungistatic drug that acts through the inhibition of the enzyme 14α-demethylase. Many dermatologists have started using higher doses and combination regimens of antifungals to counter this problem. However, such regimens have not been validated. Therefore, this study is designed to evaluate the efficacy of terbinafine and itraconazole in conventional and increased dosages and in combination in the treatment of tinea corporis, tinea cruris, and tinea faciei.

Objectives:

1. General: To evaluate the efficacy and safety of terbinafine and itraconazole in conventional and increased doses and in combination with dermatophytosis patients attending the outpatient department of Dermatology and Venereology in Dhaka Medical College Hospital.
2. Specific:

   * To evaluate the efficacy and safety of terbinafine in conventional and increased doses in dermatophytosis patients attending at the outpatient department of Dermatology and Venereology in Dhaka Medical College Hospital.
   * To evaluate the efficacy and safety of itraconazole in conventional and increased doses in dermatophytosis patients attending at the outpatient department of Dermatology and Venereology in Dhaka Medical College Hospital.
   * To evaluate the efficacy and safety of terbinafine and itraconazole in combination with dermatophytosis patients attending at the outpatient department of Dermatology and Venereology in Dhaka Medical College Hospital.
   * To observe the side effects of terbinafine and itraconazole in conventional and increased doses and in combination with dermatophytosis patients attending at the outpatient department of Dermatology and Venereology in Dhaka Medical College Hospital.

Methodology:

Study design: Randomized parallel-group trial. Place of study: Department of Dermatology and Venereology, Dhaka Medical College Hospital (DMCH), Dhaka Period of study: The study will be conducted over a period of six months from the approval of the protocol.

Study population: The dermatophytosis patients attending the outdoor Dermatology &Venereology department, Dhaka Medical College Hospital within the study period.

Sampling method: Simple Random sampling

Ethical Consideration:

Approval for the study will be obtained from the Ethical review committee of Dhaka medical college, Dhaka prior to the commencement of the study. The purpose of the study and its procedure, potential risks, and benefits will be explained to the patients in an easily understandable local language. All participating subjects will be assured that they would have the full right to withdraw themselves from the study at any time for any reason whatsoever and their refusal to participate or withdrawal from the study would not hamper their treatment anyway. They will also be assured that all records provided by them would be kept confidential and would not be disclosed anyway except for the purpose of the study. Then informed consent will be sought from them and the patients who will voluntarily consent to participate in the study will only be included.

Sample size:

The sample size is calculated using the following formula P1 = 90 (proportion of the outcome variable of the present study) P2 = 50 (known proportion of a historical control) α = 0.05 in 5% level of significance β= 0.1 in 90% power where f (α,β) is a function of α and β, the values of which is 10.5 so, n=22.3 So, a desired sample size of 25 patients in each group was calculated considering cure rates of 50% (based on current data on the effectiveness of itraconazole in India) and 90% (proportion of the outcome variable of the present study for combination therapy of terbinafine with itraconazole), with a type I error rate of 0.05, a type II error rate of 0.1. By taking 1:1 allocation and considering the dropout rates to be 20%, the final sample size calculated is 150.

Variables to be studied:

1. Socio-Demographic variables:

   * Age
   * Sex
   * Marital status
   * Occupation
   * Residence
   * Religion
   * Family history
2. Clinical variables:

   * Sites involved
   * Global improvement grade- grade I (1-25%), grade II (26-50%), grade III (51-75%), and grade IV (76-100%)11
   * Types - tinea corporis, tinea cruris and tinea faciei
3. Laboratory variables:

   * CBC,
   * LFT,
   * RFT,
   * KOH microscopy and
   * ECG

Operational definitions:

Dermatophytosis: Dermatophytosis is a superficial infection caused by a group of fungi, dermatophytes. The infection is common worldwide with higher prevalence in tropical countries.

Tinea corporis: Tinea corporis refers to any dermatophytosis of glabrous skin except palms, soles, and the groin.

Tinea cruris: Tinea cruris is a dermatophytosis of the groin, genitalia, pubic area, and perineal and perianal skin.

Tinea faciei: Tinea faciei is a dermatophytosis of the face. BSA: Body surface area (BSA) involvement will be calculated using the ' Rule of palm '. The total palmar surface of the palm and the five digits of the patient were together taken equivalent to 1%28.

PGA: The physician's global improvement(PGA) scale: The global improvement will be graded as grade I (1-25%), grade II (26-50%), grade III (51-75%), and grade IV (76-100%) improvement in overall clinical symptoms at the end of therapy.10 Efficacy: In medicine efficacy can be defined as, the ability of an intervention (a drug or surgery) to produce the desired beneficial effect.

Safety: Drug safety refers to the frequency of treatment-emergent adverse drug effects (i.e. physical or laboratory toxicity) that could possibly be related to the drug. They emerge during treatment and were not present before treatment, or they become worse during treatment compared with the pretreatment state.

Study procedure:

Participants selection: One hundred and fifty patients fulfilling the selection criteria will be randomly allocated to five parallel treatment groups on the basis of lottery and each group will contain 30 patients (allocation ratio 1: 1: 1: 1:1). Allocation will be concealed using sequentially numbered, sealed, opaque envelopes, which will contain the allocation code written on folded paper; the envelopes will be opened after enrolment of the patients. Both random sequence generation and allocation concealment will be done by a person unrelated to the trial. Skin scrapings will be taken at enrolment.

Consent and recruitment: Witnessed, written and informed consent will be taken by the patients. All female patients of childbearing age will be advised to avoid pregnancy during treatment. The patient will be evaluated on the basis of history and clinical findings and the diagnosis will subsequently be confirmed by KOH examination.

Baseline information: Socio-demographic characteristics will be assessed in terms of gender, age, religion, occupation, marital status, and place of residence. Participants will also be asked about the history of dermatophytosis among family members. Details of involved sites at the presentation and clinical course of the lesions will be registered. Clinical examination will be performed based on visual inspection and palpation. Data on location, size, clinical presentation of the lesions, and the clinical course will be recorded. Skin lesions will be encountered during the survey and will be photographed using a digital camera on every visit. The following data will be recorded for each patient: body surface area affected, treatment given, microscopy results, and investigations at baseline.

Patients will be evaluated for the severity of clinical parameters namely itching, erythema, and scaling using the four-point scale: 0 = none, l = mild, 2 = moderate, and 3 = severe. The most severe lesion will be identified as the index lesion, from which scraping and KOH microscopy will be performed at baseline and then at follow-up visits. The investigations will be performed at baseline are LFT and ECG for itraconazole groups and LFT and CBC in the terbinafine group. RFT will be done for all the groups. In combination, CBC, LFT, RFT, and ECG will be done.

Global assessment: Patients will be evaluated for the severity of clinical parameters namely itching, erythema, and scaling using the four-point scale: 0 = none, l = mild, 2 = moderate, and 3 = severe. All the patients will be followed at baseline, 2 weeks, 4, 6, and 8 weeks with repeat KOH examination from the same site, wherever necessary. The global improvement will be graded as grade I (1-25%), grade II (26-50%), grade III (51-75%), and grade IV (76-100%) improvement in overall clinical symptoms at the end of therapy.

Confidentiality: In this study, privacy, anonymity, and confidentiality of data information identifying any patient will be maintained strictly. Data taken from the participants will be coded and regarded as confidential and will be kept locked under the investigator for purposeful use only.

Participant timeline: six months.

Intervention: Five parallel study groups will be as follows:

1. Terbinafine 250 mg/day: T 1
2. Itraconazole 200 mg/day: I 1
3. Terbinafine 250 mg + Itraconazole 200 mg/day: T + I
4. Terbinafine 500 mg/day in two divided doses: T 2
5. Itraconazole 400 mg/day in two divided doses: I 2

Systemic drugs:

Patients will be prescribed the allocated antifungal drug. The same brand of drugs will be given to all the patients to rule out inter-brand variability in the efficacy of treatment. Patients will receive antihistamines (fexofenadine 180 mg). Patients will be asked to bring used strips of medicines and those in use at each visit. They will be reminded to take the medicines as prescribed at each visit and receive the treatment for 2 weeks. Patients will be advised against using any other treatment.

Topical therapy: Topical antifungals will not be prescribed. Emollient will be given to all participants.

Adherence: Adherence will be recorded in a treatment diary, which will act as an aide memoir to inform hospital appointments. Additional training will be provided at the hospital visit if it is noticed the participant will misunderstand the treatment schedule.

Follow-up: The enrolled patients will be called for follow-up every two weeks for a total of eight weeks. The following data will be recorded for each patient: body surface area affected, PGA, treatment given, microscopy results, investigations at baseline and subsequent follow-ups, and follow-up data. Investigations will be done at every second visit, LFT and ECG will be repeated in the itraconazole groups, and LFT and CBC in the terbinafine group. RFT will be done at every second visit for all the groups. In the combination group, LFT, CBC, and ECG will be repeated at every second visit. The most severe lesion will be identified as the index lesion, from which scraping and KOH microscopy will be performed at baseline and then at follow-up visits. Patients who will fail to follow up for two consecutive visits will be considered as being lost to follow-up and will be treated as dropouts.

Treatment modification following clinical response or adverse effects:

At the end of 4 weeks, those who will show no or less than 25% clinical improvement (global improvement grade I) will be labeled as 'complete failures' and will be given alternative treatment (any treatment from the rest four options); while those with partial clinical response (global improvement grades II and III) will be asked to continue same treatment for subsequent 4 weeks. if any side effects occur at any point of the treatment period then treatment will be continued with the alternate drug.

Data collection and management: Permission will be taken from each volunteer participant by using a written consent form. After getting consent from the participants, a standard questionnaire data sheet will be used to collect demographic information. The patients will be interviewed face to face by the researcher for the purpose of collection of data. All the individual's study will be subjected to a complete assessment of history and clinical examination including clinical parameters namely itching, erythema, scaling, and body surface area involvement.

Safety evaluation: All adverse events (AEs) will be assessed for severity and relationship to terbinafine and itraconazole at each visit. Multiple occurrences of the same AE will be only counted once for each patient. Laboratory measurements will also be included for safety evaluation.

Withdrawal of study participants: Each patient will enjoy every right to participate or refuse or even withdraw from the study at any point in time.

Storage: Drugs will be stored at room temperature. Prohibited medications: Any intervention for dermatophytosis, besides those provided in the trial, will be specifically prohibited.

Statistical analysis: A parametric one-way analysis of variance (F test) will be applied to find out the mean differences among the five treatment groups. The chi-square test will be used to find out significant differences in the proportions among treatment groups and it will be also used to test the significance of the change from baseline to various follow-ups within the groups. The level of significance will be set at 5% and p< 0.05 will be considered significant. Patients who will be excluded from the study due to adverse events or loss to follow-up will not be included in the data for statistical analysis.

Quality assurance strategy: In order to ensure the proper quality of the data collection procedure, firstly a work manual was made. Then a sample size was selected. A standard questionnaire was made. Then the questionnaire was 16 pretested. The pretest ensures that the respondents are able to understand the questionnaire and answer accordingly.

Utilization of results: The data generated from this study may be helpful for dermatologists to evaluate dermatophytosis treatment. Additionally, the findings of the proposed study may serve as a baseline. Data to undertake further research on a large scale.

Facilities: Resources, equipment, subjects (human), etc. required for the study]: All facilities are available in Dhaka Medical College Hospital, Dhaka. No additional facilities will be needed.

Observation and results: The result of the study and statistical analysis will be presented by tables, figures, graphs, diagrams, charts, photographs, etc. All these should have their own legends (i.e., title) and be serially numbered.

Discussion: Discussion will be done on the basis of the results obtained from the study.

Conclusion: A conclusion will be drawn depending on the results and discussion.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of tinea corporis, tinea cruris or tinea faciei or any combination of these conditions
* Microscopic confirmation of tinea (KOH microscopy showing regularly septate branching hyphae),
* Age 18- 60 years

Exclusion Criteria:

* Children less than 18 years of age
* Pregnancy and lactation
* Patients with co-existent tinea unguium, tinea pedis, or tinea manuum,
* History of recent use of antifungal drugs or steroids in last 4 weeks.
* Patient with any other disease requiring systemic therapy
* Patients with co-morbidities like cardiac disorder, liver disorder, renal disorder
* History of a drug reaction or allergy to any of the two drugs
* Any significant abnormality in complete blood counts (CBC), liver function test (LFT), renal function test (RFT), and electrocardiogram (ECG),
* Patients or attendants refused to give informed consent to take part in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of clinical parameters (itching, erythema, and scaling) | 8 weeks
  Patients will be evaluated for the severity of clinical parameters namely itching, erythema, and scaling using four-point scale as: 0 = none, l = mild, 2 = moderate, and 3 = severe. Erythema and scaling grade '0' and itching grade 0 or 1 will be considered as clinical cure.
Achievement of mycological cure at 2 weeks | 2 weeks
  Dermatophytes or yeast seen on a KOH test indicates the person has a fungal infection. The health care provider scrapes the problem area of your skin using a needle or scalpel blade. The scrapings from the skin are placed on a microscope slide. Liquid containing the chemical potassium hydroxide (KOH) is added. The slide is then examined under the microscope. A KOH examination will be done at 2 weeks and will be noted as positive or negative.
Achievement of mycological cure at 4 weeks | 4 weeks
  Dermatophytes or yeast seen on a KOH test indicates the person has a fungal infection. The health care provider scrapes the problem area of your skin using a needle or scalpel blade. The scrapings from the skin are placed on a microscope slide. Liquid containing the chemical potassium hydroxide (KOH) is added. The slide is then examined under the microscope. A KOH examination will be done at 4 weeks and will be noted as positive or negative.
Achievement of mycological cure at 6 weeks | 6 weeks
  Dermatophytes or yeast seen on a KOH test indicates the person has a fungal infection. The health care provider scrapes the problem area of your skin using a needle or scalpel blade. The scrapings from the skin are placed on a microscope slide. Liquid containing the chemical potassium hydroxide (KOH) is added. The slide is then examined under the microscope. A KOH examination will be done at 6 weeks and will be noted as positive or negative.
Achievement of mycological cure at 8 weeks | 8 weeks
  Dermatophytes or yeast seen on a KOH test indicates the person has a fungal infection. The health care provider scrapes the problem area of your skin using a needle or scalpel blade. The scrapings from the skin are placed on a microscope slide. Liquid containing the chemical potassium hydroxide (KOH) is added. The slide is then examined under the microscope. A KOH examination will be done at 8 weeks and will be noted as positive or negative.
Assessment of overall clinical symptoms with PGA | At 8 weeks
  The physician's global improvement(PGA) scale: The global improvement will be graded as grade I (1-25%), grade II (26-50%), grade III (51-75%), and grade IV (76-100%) improvement in overall clinical symptoms at the end of therapy at 8week.

SECONDARY OUTCOMES:
Assessment of treatment failure | 8 weeks
  Any of the following will be considered as treatment failure:
  * no improvement or worsening of the disease after 4 weeks in the patient's assessment,
  * the presence of scaling and/or erythema at 8 weeks, and
  * positive microscopy at 8 weeks
Patient's Satisfaction with treatment | 8 weeks
  Patients who will be cured will be asked whether they were fully satisfied with the treatment outcome or not with a yes and no answer.

IPD SHARING:
Plan to Share IPD: No